CLINICAL TRIAL: NCT05223205
Title: Optical Coherence Tomography Angiography (AngioVue™, Optovue Inc., Fremont, Calif., USA) Characteristics of Patients With Surgically Closed Full-thickness Idiopathic Macular Holes < 600 μm With Air Versus 10% SF6 Tamponade - a Pilot Study
Brief Title: Optical Coherence Tomography Angiography Characteristics of Patients With Surgically Closed Full-thickness Idiopathic Macular Holes < 600 μm With Air Versus 10% SF6 Tamponade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32-465 ex 19/20
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Macular Holes; Optical Coherence Tomography
MeSH Terms: conditions — Retinal Perforations | interventions — Air

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air group (Experimental): Air tamponade after vitrectomy.
  Interventions: Procedure: Air
- SF6 group (Experimental): 10% SF6 tamponade after vitrectomy.
  Interventions: Procedure: 10% SF6 and 90% air

INTERVENTIONS:
Procedure: Air — Test if air is sufficient for macular hole closure.
  Arms: Air group
Procedure: 10% SF6 and 90% air — Test if 10% SF6 and 90% air is sufficient for macular hole closure.
  Arms: SF6 group

SUMMARY:
State of the art treatment for idiopathic macular holes consists of pars plana vitrectomy, internal limiting membrane staining with a blue colouring dye, internal limiting membrane peeling and filling of the vitrectomized space with a specific tamponade such as air and SF6. Air and SF6 have previously shown similar closure rates, although there was a trend towards lower closure rates in large diameter IMH (Idiopathic Macular Holes) using air. IMH with diameters < 600 μm are currently believed to have similar closure rates with air and SF6. The investigators want to assess possible effects of the used tamponade (air or SF6) on closure rates and perfusion parameters represented by OCTA (Optical coherence tomography angiography). IMH eyes with a minimum diameter > 600 μm will be excluded. Two idiopathic macular hole patient groups will therefore be formed: The first group (group 1) will receive air after vitrectomy and membrane peeling, the second group (group 2) will receive 10% SF6 (and 90% air) after vitrectomy and membrane peeling. After recruitment, patients will therefore be electronically randomized to one of the two groups. The groups will then be compared by the means of OCT (Optical coherence tomography) and OCTA.

Note: The trial was registered retrospectively on Clinicaltrials.gov after start of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able and willing to give informed consent.
* Patient must be between 18 and 100 years of age.
* Patient must not have any significant media opacity which interferes with the examination.
* Patient must have an (stage 1-4) idiopathic macular hole requiring surgery.

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Under 18 or over 100 years of age
* Significant media opacities
* Systemic pathologies making an examination difficult or cumbersome to the patient
* Primary and/or secondary epiretinal membranes (ERM), except incipient ERMs not affecting the foveal contour and not requiring surgery
* Full-thickness idiopathic macular hole > 600 μm in minimum diameter
* Nonclosure
* Lamellar holes not requiring surgery
* Pseudo holes
* Glaucoma
* Diabetes
* Anisometropia > 2 diopters
* High myopia (spherical equivalent > 6 diopters and/or axial length > 26 mm
* Other retinal or ophthalmic pathologies except moderate cataract
* OCTA scan signal strength < 5
* Low image quality
* Failure of automatic layer segmentation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Macular hole closure | 2 weeks

SECONDARY OUTCOMES:
Foveal avascular zone area | 3 months
Parafoveal vessel density | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided